CLINICAL TRIAL: NCT01434251
Title: Treatment of Hypotension of Prematurity: a Randomized, Non-blinded Cohort Clinical Trial
Brief Title: Treatment of Hypotension of Prematurity (TOHOP)
Acronym: TOHOP
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: It was decided to conclude recruitment due to declining eligibility/recruitment rates and an unrealistically long time span to reach full recruitment.
Sponsor: UMC Utrecht (Other)
Responsible Party: Principal Investigator, Petra Lemmers, MD PhD, UMC Utrecht
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: NL 33865.041.10
Record Dates: First submitted 2011-09-09; First posted 2011-09-14 (Estimated); Last update posted 2024-12-16 (Actual); Status verified 2024-12

CONDITIONS: Hypotension
Keywords: Hypotension; premature infants; near infrared spectroscopy
MeSH Terms: conditions — Hypotension; Premature Birth

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Standard care (Active Comparator): Infants will be treated according to the treatment policy operative in the Neonatal Intensive Care Unit (NICU) of the Wilhelmina Children's Hospital/University Medical Centre Utrecht (UMCU): anti-hypotensive therapy will be started when the mean blood pressure (in mmHg) is below the gestational age in weeks.
  Interventions: Other: Anti-hypotensive treatment
- Delayed intervention (Other): Anti hypotensive therapy will be started when the mean blood pressure (in mmHg) is < (gestational age in weeks - 5 mmHg) or when there is clinical or biochemical evidence of impaired tissue perfusion.
  Interventions: Other: Anti-hypotensive treatment

INTERVENTIONS:
Other: Anti-hypotensive treatment — Hypotension is managed using a variety of treatment options. Options include: fluid bolus(es), dopamine, dobutamine, hydrocortisone and epinephrine.

SUMMARY:
Hypotension in the very preterm infant (gestational age [GA] <32 wks) is a frequently occurring clinical problem. Although no real consensus has been reached on the definition of hypotension in these infants, in clinical practice a mean blood pressure (mean BP) in mmHg lower than the GA age in weeks is considered to be the starting point for anti-hypotensive therapy. However, although an association between neonatal hypotension and mortality/ morbidity exists, there is no evidence of causality between hypotension (meanBP <GA in completed weeks) and neonatal mortality/morbidity. In addition, using mean BP alone as the indication of treatment of neonatal cardiovascular compromise without taking into consideration the status of tissue perfusion may lead to unnecessary exposure of neonates to vasoactive medication. This medication can be potentially harmful to these extremely vulnerable patients.

The aim of this study is to compare neonatal mortality and short-term neurodevelopmental outcome (cerebral ultrasound during the first 7 days of life, advanced MRI indices of structural brain injury at term GA) and long-term neurodevelopmental outcomes (Bayley scales of infant development III [BSID-III] at 24 months) between two groups of very preterm infants presenting with hypotension without clinical and laboratory evidence of compromised tissue perfusion during the first 3 days of life. Hypotension will be defined as the mean BP (in mm Hg) lower than the infant's GA (in weeks). Patients randomized to "Group A" will be treated according to the treatment protocol operative in the Neonatal Intensive Care Unit (NICU) of the University Medical Centre Utrecht (UMCU) while "Group B" will receive no cardiovascular support for hypotension unless they have evidence of compromised tissue perfusion and end-organ function ((i.e. near infrared-monitored regional cerebral oxygen saturation (ScO2) <50% despite optimized ventilatory support and FiO2 administration, plasma lactate >6 mmol/L; and/or urine output <0.6 mL/kg/hour) or mean BP >5mmHg lower than the current guideline.

The investigators hypothesize that there will be no differences between the two groups concerning short and long-term neurodevelopmental outcomes.

DETAILED DESCRIPTION:
Rationale: Hypotension in the very preterm infant (gestational age [GA] <32wks) is a frequently occurring clinical problem. Although no real consensus has been reached on the definition of hypotension in the very preterm baby, in clinical practice a mean blood pressure (BP) in mmHg lower than the GA age in weeks is considered to be the starting point for anti-hypotensive therapy. However, although an association between neonatal hypotension and mortality and morbidity exists, there is no evidence of causation between hypotension and neonatal mortality and morbidity (including neurodevelopmental outcome at 2 and 3 years of age). In addition, using mean BP alone as the indication of treatment of neonatal cardiovascular compromise without taking into consideration information on the status of tissue perfusion may lead to unnecessary exposure of neonates to forceful vasoactive medications potentially causing harm to these extremely vulnerable patients.

Objective: To compare neonatal mortality and short-term (advanced MRI indices of structural brain injury at 40 weeks' GA) and long-term neurodevelopmental outcomes (Bayley scales of infant development III [BSID-III] at 24 months) between two groups of very preterm infants presenting with hypotension without clinical and laboratory evidence of compromised tissue perfusion during the first 72 postnatal hours (3 days). Hypotension will be defined as the mean BP (in mm Hg) lower than the infant's GA (in weeks). Patients randomized to "Group A" will be treated according to the treatment policy operative in the Neonatal Intensive Care Unit (NICU) of the Wilhelmina Children's Hospital/University Medical Centre Utrecht (UMCU) while "Group B" will receive no cardiovascular support for hypotension unless they have a mean BP lower than the current limit minus 5 mmHg and/or evidence of compromised tissue perfusion and end-organ function and thus meet established criteria (see below).

Study design: A single-centre randomized non-blinded cohort study in the NICU at the UMCU of preterm neonates <30 weeks' gestation during postnatal days 0 to 3.

Study population: All preterm infants with a GA of <30 weeks admitted on day of postnatal life 0 to the NICU at the UMCU. Patients will be managed according to their randomization to Group A or B until the end of postnatal day 3.

Intervention Patients randomized to "Group A" will be treated for hypotension according to the treatment protocol operative in the NICU at the UMCU. Patients randomized to "Group B" will receive no cardiovascular supportive therapy irrespective of their BP value unless their mean BP is >5 mmHg below GA in weeks for 30 minutes and/or they have indirect clinical or direct laboratory evidence of tissue hypoperfusion and/or end-organ dysfunction (i.e. rScO2 is <50% despite optimized ventilatory support and FiO2 administration, plasma lactate >6 mmol/L; and/or urine output <0.6 mL/kg/hour).

As CO2 is the most potent regulator of cerebral blood flow (CBF), it is understandable why changes in arterial CO2 tension (PaCO2) has been associated with increased incidence of peri-intraventricular hemorrhage (PIVH) in preterm neonates with significant hypercapnia and with white matter injury (periventricular leukomalacia; PVL) in preterm neonates with hypocapnia during the immediate postnatal period. Therefore, in the present study, ventilation will be closely followed and PaCO2 values monitored and attempted to be kept within normal limits (40-to-50 mmHg) during the first three postnatal days to control for the potential impact of this confounding variable as far as the primary and secondary outcome measures are concerned (see below).

Main study parameters/endpoints: To determine whether refraining (group B) from anti-hypotensive treatment has a negative, positive or no effect on the composite outcome of mortality and neurodevelopmental outcome (determined by BSID-III) at 24 months of age. Secondary outcome measures will include 1) differences between the groups in the incidence of PIVH during the first 7 postnatal days detected by head ultrasound, 2) differences in the incidence of white matter injury PVL and gray matter injury not detected within the first 7 days by ultrasound using advanced MRI parameters of the brain at the adjusted postmenstrual age of 40 weeks as well as the ability to maintain CBF autoregulation during the first three postnatal days.

ELIGIBILITY:
Inclusion Criteria:

* Idiopathic arterial hypotension as defined by a mean BP in mmHg less than the GA in weeks at birth.
* Written parental consent

Exclusion Criteria:

* Prior inclusion indirect clinical or direct laboratory evidence of poor organ/tissue perfusion (plasma lactate >6 mmol/L on two consecutive measurements and/or urine production <0.6 mL/kg/h for a 6-hour period
* Clinically and/or microbiologically proven sepsis
* Major congenital abnormalities
* Postnatal age at the time of the development of systemic hypotension >72 hours
* No arterial line for continuously monitoring of blood pressure

Ages: 24 Weeks to 30 Weeks | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 150 (Estimated)
Dates: Start 2011-09-01 (Actual); Primary Completion 2021-02-01 (Actual); Study Completion 2021-02-01 (Actual)

PRIMARY OUTCOMES:
Neurodevelopmental outcome assessment using the Bayley Scales of Infant Development III | 24 months postnatal age.

SECONDARY OUTCOMES:
Incidence of peri-intraventricular haemorrhage | first 7 postnatal days.
  As detected by cranial ultrasound
Incidence of white matter injury and gray matter injury | adjusted postmenstrual age of 40 weeks
  White/gray matter injury assessed by using advanced MRI indices.
Difference in the ability to maintain cerebral blood flow autoregulation | Determined from start of hypotensive period (expected within 24h postnatal age) until end of hypotensive period (expected average of 72h postnatal age)
  Assessed by determining the correlation between the mean arterial blood pressure and cerebral oxygenation (rScO2).
Mortality | Duration of follow-up (24 months postnatal age)

CONTACTS AND LOCATIONS:
Overall Officials: Petra MA Lemmers, MD, PhD, Principal Investigator — UMC Utrecht; Thomas Alderliesten, MD, Principal Investigator — UMC Utrecht
Locations (1):
- Wilhemlina Childrens Hostpital/University Medical Center Utrecht, Utrecht, Utrecht, Netherlands

REFERENCES:
- [Derived] Alderliesten T, Arasteh E, van Alphen A, Groenendaal F, Dudink J, Benders MJ, van Bel F, Lemmers P. Treatment of Hypotension of Prematurity: a randomised trial. Arch Dis Child Fetal Neonatal Ed. 2025 Dec 15;111(1):F60-F66. doi: 10.1136/archdischild-2024-328253. PMID 40413017